CLINICAL TRIAL: NCT02739958
Title: Effects of Propofol-dexmedetomidine on Immune Function During Total Laryngectomy Surgery Compared With Isoflurane Anesthesia
Brief Title: Effects of Propofol-dexmedetomidine on Immune Function in Patients With Cancer Larynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R/16.01.112
Record Dates: First submitted 2016-03-11; First posted 2016-04-15 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Cancer Larynx; Total Laryngectomy
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol group (Active Comparator): Patients receive only intravenous anesthetics
  Interventions: Drug: Propofol group
- Isoflurane group (Placebo Comparator): Patients receive isoflurane /fentanyl anesthesia
  Interventions: Drug: Isoflurane group

INTERVENTIONS:
Drug: Propofol group — Anesthesia is maintained with continuous infusion of propofol 1.5-2mg/kg/h and dexmedetomidine 0.2-1ug/kg/h.
  Arms: Propofol group
Drug: Isoflurane group — Anesthesia was maintained with isoflurane at a concentration of 2-2.5%. fentanyl 50 ug increments
  Arms: Isoflurane group

SUMMARY:
The aim of this prospective, randomized clinical study is to compare between propofol and isoflurane on perioperative immune cell populations and function in patients undergoing total laryngectomy surgery.

DETAILED DESCRIPTION:
The perioperative period might be a critical time in primary cancer surgery because many factors can affect whether recurrence, or metastasis , or elimination by the immune system.

Cancer surgery can induce an acute inflammatory response, due to local tissue damage and the shedding of malignant cells into the blood and lymphocytic circulation although meticulous surgical manipulation. Many evidences suggest that several factors during the perioperative period can affect the immune system.

These could be attributed to the surgery per se, pain, anxiety, hypothermia, blood transfusion, anesthetic technique, and anesthetic drugs .Impairment in the immune system may allow malignant cells to escape immuno-surveillance and metastasize in the perioperative period.As well as increase the risk of postoperative complications, such as systemic inflammatory response syndrome, sepsis, and multi-organ failure.

Previous retrospective clinical studies of both breast and prostate cancer surgery have suggested an association between anaesthetic technique and cancer recurrence.

However ,other retrospective trials on various forms of cancer have shown no such benefit.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I- III
* Scheduled for total laryngectomy.

Exclusion Criteria:

* Patients refusal.
* Morbid obese patients (body mass index >40 kg/m2).
* Allergy to local anesthetics agents used.
* Severely altered consciousness level.
* Psychiatric disorders.
* Severe or uncompensated cardiovascular disease.
* Severe renal disease.
* Severe hepatic disease.
* Severe endocrinal diseases.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
CD3 plasma level | for 7 days after procedure
  Venous blood samples will be collected. The extracted venous blood samples will be mixed evenly in a special anti-coagulation test tube and stored in a refrigerator (at 4C).Flow cytometer will be used to detect the level of CD3+

SECONDARY OUTCOMES:
Heart rate | for 5 hours during the procedure
  Intraoperative heart rate changes
Blood pressure | for 5 hours during the procedure
  Intraoperative blood pressure changes
Peripheral oxygen saturation measured with pulse oximetry | for 5 hours during the procedure
  Intraoperative peripheral oxygen saturation changes as measured with pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Reem A El Sharkawy, MD, Principal Investigator — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University Hospitals, Ear Nose Thorat Department, Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided